CLINICAL TRIAL: NCT01791374
Title: A Multicenter, Phase 1/1b, Open Label Study Evaluating the Safety, Tolerability and Pharmacokinetics of Rilotumumab in Japanese Subjects
Brief Title: Phase 1/1b Study of Rilotumumab in Japanese Subjects With Advanced Solid Tumors or Advanced or Metastatic Gastric or GEJ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110251; 20110251 (Other: Amgen)
Record Dates: First submitted 2013-01-04; First posted 2013-02-15 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Part 1- Advanced Solid Tumors; Part 2- Advanced or Metastatic Gastric Cancer; Part 2- Advanced or Metastatic GEJ
Keywords: Advanced Solid Tumors; Advanced or Metastatic Gastric Cancer; Advanced or Metastatic GEJ; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — rilotumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rilotumumab Monotherapy (Experimental): Cohort 1A: Rilotumumab 10 mg/kg IV Q2W Cohort 1B: Rilotumumab 20 mg/kg IV Q2W Cohort 1C (if needed): Rilotumumab 15 mg/kg IV Q2W
  Interventions: Drug: Rilotumumab
- Rilotumumab plus CX (Experimental): Cohort 2A: Rilotumumab 15 mg/kg IV Day 1 Q3W Cisplatin 80 mg/m2 IV (max of 6 cycles) Day 1 Q3W Capecitabine 1000 mg/m2 PO BID, Days 2-14 Q3W Cohort 2B (if needed): Rilotumumab 10 mg/kg IV Day 1 Q3W Cisplatin 80 mg/m2 IV (max of 6 cycles) Day 1 Q3W Capecitabine 1000 mg/m2 PO BID, Days 2-14 Q3W
  Interventions: Drug: Rilotumumab

INTERVENTIONS:
Drug: Rilotumumab — Rilotumumab is a fully human monoclonal antibody immunoglobulin G, type 2 (IgG2) against human hepatocyte growth factor/scatter (HGF/SF) that blocks binding of HGF/SF to its receptor MET, inhibiting HGF/MET-driven activities in cells.
  Other Names: AMG 102
  Arms: Rilotumumab Monotherapy
Drug: Rilotumumab — Drug: Rilotumumab Rilotumumab is a fully human monoclonal antibody immunoglobulin G, type 2 (IgG2) against human hepatocyte growth factor/scatter (HGF/SF) that blocks binding of HGF/SF to its receptor MET, inhibiting HGF/MET-driven activities in cells. Drug: Cisplatin A platinum containing chemo-therapy compound that reacts in vivo, binding to and causing crosslinking of DNA, which ultimately triggers apoptosis (programmed cell death). Drug: Capecitabine A chemo-therapy prodrug, that is enzymatically converted to 5-fluorouracil in the tumor, where it inhibits DNA synthesis and slows growth of tumor tissue.
  Other Names: AMG 102
  Arms: Rilotumumab plus CX

SUMMARY:
This is an open label phase 1/1b study of Rilotumumab in Japanese subjects with advanced solid tumors or metastatic gastric esphagogastric (GEJ) adenocarcinoma.

ELIGIBILITY:
Key Inclusion Criteria:

* Japanese subjects with pathologically confirmed unresectable locally advanced or metastatic carcinoma which is refractory to standard therapies or for which there is no standard therapy (Part 1 only)
* Japanese subjects with pathologically confirmed MET-positive (fulfilling the MET IHC criteria as defined by validated IVD [in vitro diagnostic]) unresectable locally advanced or metastatic gastric or GEJ adenocarcinoma (Part 2 only)
* Eastern Cooperative Oncology Group (ECOG) Performance Status (0 or 1)
* Availability of archival tumor tissue (Part 2 only)
* Evaluable (measurable or non-measurable) disease by RECIST 1.1 criteria
* Able to tolerate infusions and take oral medications (Part 2 only)

Key Exclusion Criteria:

* Previous systemic therapy (including chemotherapy, biologic, immunotherapy, or investigational therapy) for locally advanced or metstatic gastric or GEJ adenocarcinoma (Part 2 only)
* Less than 6 months have elapsed from completion of prior neoadjuvant or adjuvant chemotherapy or chemotherapy to enrollment (Part 2 only)
* Squamos cell history (Part 2 only)
* Known HER2-overexpressing unresectable locally advanced or metastatic gastric or GEJ adenocarcinoma (Part 2 only)
* Resectable disease or suitable for definitive chemoradiation
* Subjects who have persistent gastric outlet obstruction, complete dysphagia or are dependent upon jejunostomy for feeding (Part 2 only)
* Known central nervous system metastases

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Part1: Dose-limiting toxicities (DLT) for each dose level of rilotumumab tested | 28 days
  DLTs are defined as grade 3 or higher adverse events that are related to rilotumumab during the first cycle of therapy. This does not include specific toxicities (eg nausea and vomiting) that are common in cancer patients unless specific criteria are met.
Part 2: Dose-limiting toxicities (DLT) for each dose level of rilotumumab in combination with cisplatin and capecitabine (CX) chemotherapy tested | 21 days
  DLTs are defined as grade 3 or higher adverse events that are related to rilotumumab or the combination of rilotumumab and CX during the first cycle of therapy. This does not include specific toxicities (eg nausea and vomiting) that are common in cancer patients unless specific criteria are met.

SECONDARY OUTCOMES:
Part 1: Incidence of AEs, clinical laboratory abnormalities and anti-rilotumumab antibodies. | 4 months average
  AEs and laboratory abnormalities are reported by CTCAE (version 3.0) criteria
Part 1: Pharmacokinetics parameters of rilotumumab monotherapy as measured by: Maximum concentration, time to achieve maximum concentration, observed minimum concentration, area under the concentration-time curve, terminal elimination half-life. | 4 months average
Part 1: Evaluate efficacy based on the treatment effects of rilotumumab monotherapy as measured by the following: Objective Response Rate, duration of response, progression-free survival. | 4 months average
Part 2: Incidence of AEs, clinical laboratory abnormalities and anti-rilotumumab antibodies not defined as DLTs. | 7 months average
  AEs and laboratory abnormalities are reported by CTCAE (version 3.0) criteria
Part 2: Pharmacokinetics parameters of rilotumumab in combination with cisplatin and capecitabine as measured by: Maximum concentration, observed minimum concentration, area under the concentration-time curve. | 7 months average
Part 2: Evaluate efficacy based on the treatment effects of rilotumumab in combination with cisplatin and capecitabine as measured by the following: Objective Response Rate, duration of response, progression-free survival, overall survival. | 7 months average

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- Japan (7):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Kashiwa-shi, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Kitaadachi-gun, Saitama
  - Research Site, Suntou-gun, Shizuoka

REFERENCES:
- [Derived] Doi T, Yamaguchi K, Komatsu Y, Muro K, Nishina T, Nakajima TE, Tang R, Yang H, Zhang Y, Jung AS, Ang A, Yasui H. A Phase 1/1b tolerability study of rilotumumab alone or in combination with cisplatin and capecitabine in Japanese patients with gastric cancer. Jpn J Clin Oncol. 2017 Nov 1;47(11):1002-1009. doi: 10.1093/jjco/hyx114. PMID 28973403
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com